CLINICAL TRIAL: NCT04162496
Title: An Evaluator -Blinded, Split-Neck, Randomized Clinical Study Investigating the Efficacy and Safety of Restylane Refyne for Correction of Static Horizontal Neck Rhytides Utilizing Either a Cannula or Needle
Brief Title: Restylane Refyne for Correction of Horizontal Neck Rhytides
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siperstein Dermatology (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Robyn Siperstein, Primary Investigator, Siperstein Dermatology
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SipDerm
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Aging; Wrinkle; Rhytides
Keywords: Hyaluronic Acid Filler; Neck Rhytides; Transverse Neck Lines; Tech Neck; Necklace Lines; Restylane; Restylane Refyne

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment with Restylane Refyne Group 1 (Experimental): Treat right side with Restylane Refyne with a cannula and left side with a needle
  Interventions: Device: Restylane Refyne
- Treatment with Restylane Refyne Group 2 (Experimental): Treat left side with Restylane Refyne with a cannula and right side with a needle
  Interventions: Device: Restylane Refyne

INTERVENTIONS:
Device: Restylane Refyne — Injection of Restylane Refyne with a cannula on one side of the neck and a 30 guage needle on the other side.

SUMMARY:
Subjects with grades ranging from 1---3 on the Transverse Neck Line Scale, will be randomized to receive up to 1cc of Restylane Refyne on one side of their neck utilizing a cannula and up to 1cc of Restylane Refyne on the other side utilizing a 30--gauge needle. On Day 30, this treatment with the same left---right assignment can be repeated if optimal correction on either side has not been achieved according to the treating investigator. Subjects will return 24--48 hours after their first treatment, to fill out questionnaires, take pictures, and to be assessed by blinded evaluators regarding adverse events. Subjects will also return 30 days after their final treatment to fill out final questionnaires, take pictures, and to be assessed by blinded evaluators regarding improvement of static rhytides.

DETAILED DESCRIPTION:
This will be a prospective, evaluator-blinded, split--neck, clinical study in which patients will be randomized to 2 groups.

The first group will receive up to 1cc of Restylane Refyne into the rhytides on the right side of the neck utilizing a 27---gauge cannula, while the left side will be injected with a sharp 30--gauge needle.

The second group will be reversed with the left side treated with Restylane Refyne utilizing a cannula and the right side treated with a sharp needle.

Both groups will be utilizing the same safety and comfort protocols established by the practice which include the use of topical numbing cream (B.L.T.), cleansing with alcohol, and a cold ice pack at the site of injection after the procedure.

Before and after the procedure a set of blinded evaluators will be grading the subjects' static horizontal neck lines using a validated 5--point grading scale. The blinded evaluators will also be grading the subjects side effects such as bruising and swelling 24---48 hours after the first treatment. A second treatment is allowed on Day 30 for those who have not achieved optimal correction. Either on Day 30 or Day 60, a final assessment with digital photography using Canfield's Vectra imaging system, along with a patient questionnaire on satisfaction, improvement (GAIS), side effects, and pain levels during and after the procedure will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* In good general health as evidenced by medical history
* For females of reproductive potential: use of highly effective contraception
* Score of 1--3 on a validated transverse neck line scale3

Exclusion Criteria:

* Subjects with allergies to hyaluronic acid filler.
* Subjects with auto--immune conditions
* Subjects with diabetes
* Subjects taking anti--coagulants, diuretics, anti-histamines, or anti--inflammatory medications in the 2 weeks prior to the study or who will need to take these medications at any time during the 60 day study.
* Subjects with any scheduled laser, light, or surgical procedures during the study, including dental surgery.
* Subjects who had neuromodulators in the past 6 months or fillers in the previous 2 years in the neck area
* Subjects who at any time had surgery or permanent fillers in the neck area
* Subjects with scars, tattoos, or many skin growths in the neck area
* Subjects unwilling or unable to sit still while an injector places Restylane Refyne in the neck
* Subjects unwilling or unable to keep their head still during the photos
* Subjects who are pregnant or nursing
* Female subjects unable to take or use some form of birth control
* Subjects with any neck bruising or swelling
* Subjects with current skin infections, tumors, herpes outbreak or dermatitis on the neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in transverse neck rhytides | Baseline to 30 days after the last treament
  Difference in the mean absolute change from baseline on a 5--point validated transverse neck line scale. The lowest score 0 signifies no line and a better outcome while the highest score 4 signifies a worse outcome.

SECONDARY OUTCOMES:
Adverse Events | Day 1 to Day 30
  The number of reported adverse events and the difference between the two sides in the mean number of adverse events
Global Aesthetic Improvement Scale | 30 Days after the last treatment
  Global aesthetic improvement scale as rated by subjects and evaluators. This is a 4 point scale with a 5 point scale with a -1 as the lowest score signifying a lower outcome and 3 as the highest score signifying the best outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Siperstein Dermatology, Boynton Beach, Florida, United States